CLINICAL TRIAL: NCT03919084
Title: A Pharmacy Liaison-Patient Navigation Intervention to Reduce Inpatient and Emergency Department Utilization Among Primary Care Patients in a Medicaid Accountable Care Organization: A Pragmatic Trial
Brief Title: THRIVE+ Pharmacy Liaison-Patient Navigation Intervention
Acronym: THRIVE+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Massachusetts Health Policy Commission (Other); John Hancock Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-38000
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Healthcare Utilization
Keywords: THRIVE; Patient navigation; Accountable Care Organization; Pharmacy liaison; Pharmacy services; Social determinants of health; health-related social needs; screening and referral; Medicaid ACO; ACO
MeSH Terms: interventions — Referral and Consultation; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE-Basic (Active Comparator): Screening-and-referral usual care model
  Interventions: Other: THRIVE screening and referral; Other: Pharmacy Care Program services
- THRIVE+ (Experimental): Enhanced screening-and-referral with motivational interviewing and patient navigation services
  Interventions: Other: THRIVE screening and referral; Other: Pharmacy Care Program services; Other: Patient Navigation Services; Other: Motivational Interviewing; Other: Linkage to Community Partner Organization

INTERVENTIONS:
Other: THRIVE screening and referral — The THRIVE screening tool includes questions to identify eight potentially unmet health-related social needs associated with health outcomes and healthcare utilization: housing and food insecurity, inability to afford medications, need for transportation, trouble paying for heat and electricity, need for employment or education, and difficulty taking care of children or other family members. The survey is written at a 3rd grade reading level, is available in multiple languages, and requires less than five minutes to complete. The paper screener consists of two parts: part one screens patients for health-related social needs in the eight domains. Part two asks patients to indicate the resources they want help accessing across the eight domains. Patients who request resources in one or more domains receive paper guides that describe available hospital and community resources to address the specific domain(s) indicated.
  Other Names: THRIVE-Basic
Other: Pharmacy Care Program services — Pharmacy services provided by a pharmacy liaison include assessing gaps in obtaining refills, identifying barriers to medication adherence, reviewing the patient's engagement in medical care, and developing an action plan with the patient. Action plans focus on strategies to increase medication adherence and engagement in care. The pharmacy liaison will also link the patient to a clinical pharmacist, when appropriate, and will assist the patient with prescription management. After the initial intake is completed, the pharmacy liaison will call patients monthly (or meet with them prior to or following scheduled appointments) over a twelve-month period to confirm medication adherence and address any new barriers to medication adherence and engagement in medical care. The pharmacy liaison in the control arm does not systematically initiate screening for health-related social needs.
Other: Patient Navigation Services — In traditional patient navigation programs, a lay person from the community guides individuals through the healthcare system to receive appropriate services. For the present study, the research team will train pharmacy liaisons (pharmacy technicians or pharmacy interns with at least a high school degree and four years of pharmacy experience) to provide patient navigation services, in addition to providing medication adherence support and assistance resolving barriers to accessing medication. In an effort to avoid duplication of services the patient navigation intervention will be delivered via a pharmacy liaison trained in patient navigation, thereby decreasing multiple intervention providers and increasing the potential for sustainability should the intervention prove effective.
  Arms: THRIVE+
Other: Motivational Interviewing — Motivational interviewing is a counseling method that encourages patient-centered discussions. Motivational interviewing will be delivered by the intervention arm pharmacy liaison-patient navigators to identify the patient's unmet needs and encourage the patient to adopt behavior change that will promote engagement with resources and services to mitigate or alleviate HRSN.
  Arms: THRIVE+
Other: Linkage to Community Partner Organization — The pharmacy liaison-patient navigator will partner with a community organization, Action for Boston Community Development (ABCD). ABCD will help connect patients receiving THRIVE+ to community resources including childcare, food, heating, and housing. The pharmacy liaison-patient navigator will interface directly with ABCD to coordinate receipt of resources for their patients.
  Arms: THRIVE+

SUMMARY:
This is a pragmatic comparative effectiveness trial (n=364) to compare two screening and referral program models to address health-related social needs (HRSN) among the intermediate risk population of Boston Accountable Care Organization (BACO), a Medicaid ACO. The first study arm is THRIVE-Basic, the low-touch usual care model already implemented in all primary care clinics at Boston Medical Center (BMC) where patients are screened for HRSN and receive a printed paper resource referral guide. The second study arm is THRIVE+, which enhances the THRIVE-Basic model by engaging a pharmacy liaison-patient navigator to provide targeted navigation services and motivational interviewing to ensure connection to hospital- and community-based resources. The patient navigators will also interface directly with a partner community organization, Action for Boston Community Development (ABCD), to further help connect patients receiving THRIVE+ to community resources for HRSN. All patients in our study will receive pharmacy services via an existing Pharmacy Care Program. Patients in study arm 1 will be connected to a pharmacy liaison, which is standard clinical practice for intermediate risk ACO members in the BMC General Internal Medicine clinics. Patients in study arm 2 will receive systematic screening for and addressing of HRSN (THRIVE+) via a pharmacy liaison-patient navigator (a pharmacy technician trained as a patient navigator to deploy both pharmacy services and the THRIVE+ intervention), thereby avoiding duplication of services and multiple touches. Assignment to the study arms will be linked to existing Pharmacy Care Program enrollment activities and will be based on medical record number. The investigators' rationale for the study is that if patients' HRSN are addressed, patients will be better positioned to manage chronic conditions, adhere to preventive care plans, and less likely to use the emergency department (a conduit to inpatient care) for ambulatory care-sensitive conditions. The effectiveness of these two models will be compared with respect to alleviating HRSN and reducing acute health care utilization over a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Identified as within the 3rd to 10th percentile for healthcare utilization and cost among Boston Accountable Care Organization (BACO) Medicaid ACO membership at the time of enrollment in the clinical program; and
* Attend a primary care visit with a primary care provider (PCP-nurse practitioner or physician) in General Internal Medicine at Boston University Medical Center.

Exclusion Criteria:

-Patients who are receiving services from the BACO complex care management program.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 364 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2021-03-05 (Actual); Study Completion 2021-03-05 (Actual)

PRIMARY OUTCOMES:
Acute healthcare utilization composite measure | 12 months
  Measure includes all-cause hospital admissions and all-cause emergency department visits.

SECONDARY OUTCOMES:
Number of all-cause emergency department visits | 12 months
  Total number of all-cause emergency department visits.
Number of 30-day emergency department revisits | 12 months
  Total number of all-cause emergency department revisits within thirty (30) days of initial emergency department visit.
Emergency department revisits rate | 12 months
  Total number of all-cause emergency department revisits within thirty (30) days of initial emergency department visit divided by total number of all-cause emergency department visits.
Number of all-cause hospital discharges | 12 months
  Total number of all-cause discharges from inpatient status
Number of 30-day hospital readmissions | 12 months
  Total number of all-cause discharges from inpatient status that had a subsequent admission within thirty (30) days of the initial discharge.
30-day inpatient readmission rate | 12 months
  Total number of all-cause discharges from inpatient status that had a subsequent admission within thirty (30) days of the initial discharge divided by total number of all-cause discharges from inpatient status.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Lasser, MD MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buitron de la Vega P, Ashe EM, Xuan Z, Gast V, Saint-Phard T, Brody-Fialkin J, Okonkwo F, Power J, Wang N, Lyons C, Silverstein M, Lasser KE. A Pharmacy Liaison-Patient Navigation Intervention to Reduce Inpatient and Emergency Department Utilization Among Primary Care Patients in a Medicaid Accountable Care Organization: A Nonrandomized Controlled Trial. JAMA Netw Open. 2023 Jan 3;6(1):e2250004. doi: 10.1001/jamanetworkopen.2022.50004. PMID 36622674
- [Derived] Lasser KE, Buitron de la Vega P, Ashe EM, Xuan Z, Alva S, Battisti L, Losi S, Sieber C, Richards C, Sullivan P, Triscari L, Brody L, Roth MT, LeBlanc A, Silverstein M. A pharmacy liaison-patient navigation intervention to reduce inpatient and emergency department utilization among primary care patients in a Medicaid accountable care organization: A pragmatic trial protocol. Contemp Clin Trials. 2020 Jul;94:106046. doi: 10.1016/j.cct.2020.106046. Epub 2020 May 31. PMID 32485325